CLINICAL TRIAL: NCT00744978
Title: A Phase 2 Multicenter, Double-Blind, Placebo-Controlled, Crossover Trial of Varenicline Tartrate (CP-526,555) in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Evaluation of the Efficacy of Varenicline on Cognition, Safety, Tolerability and Pharmacokinetics in Subjects With Mild-to-Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A3051101
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Results first posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-10

CONDITIONS: Alzheimer's Disease
Keywords: Efficacy; Safety; Pharmacokinetics; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Experimental)
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — 0.5 mg once daily for 1 week followed by 0.5 mg twice daily for 1 week followed by 1 mg twice daily for 4 weeks
  Other Names: Chantix, Champix
  Arms: Varenicline
Drug: Placebo — Placebo once daily for 1 week followed by placebo twice daily for 5 weeks.
  Arms: Placebo

SUMMARY:
1. Assess the efficacy of varenicline, relative to placebo, on a performance based measure of cognition in patients with mild to moderate Alzheimer's disease
2. Evaluate the effects of varenicline on clinically relevant measures including attention and executive function, behavior, and clinician rated global change.
3. Evaluate the safety and tolerability of varenicline, relative to placebo, in patients with mild to moderate Alzheimer's disease
4. Evaluate the pharmacokinetics of varenicline in patients with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, age 55-85
* Diagnosis of probable Alzheimer's disease, consistent with criteria from both: 1) National Institute of Neurological and Communicable Disease and Stroke and Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) and 2) Diagnostic and Statistical Manual of Mental Disorders (DSM IV)
* Mini-mental status exam score of 14-26 inclusive
* Rosen-Modified Hachinski Ischemia Score of < or = 4

Exclusion Criteria:

* Diagnosis or history of other dementia or neurodegenerative disorders
* Diagnosis or history of clinically significant cerebrovascular or cardiovascular disease
* Subjects with pulmonary disease or evidence of clinically significant pulmonary symptoms

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- South Korea (6):
  - Pfizer Investigational Site, Seongnam, Gyunggido
  - Pfizer Investigational Site, Busan
  - Pfizer Investigational Site, Daegu
  - Pfizer Investigational Site, Incheon
  - Pfizer Investigational Site, Seoul
  - Pfizer Investigational Site, Suwon

REFERENCES:
- [Derived] Kim SY, Choi SH, Rollema H, Schwam EM, McRae T, Dubrava S, Jacobsen J. Phase II crossover trial of varenicline in mild-to-moderate Alzheimer's disease. Dement Geriatr Cogn Disord. 2014;37(3-4):232-45. doi: 10.1159/000355373. Epub 2013 Nov 14. PMID 24247022
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051101&StudyName=Evaluation%20of%20the%20Efficacy%20of%20Varenicline%20on%20Cognition%2C%20Safety%2C%20Tolerability%20and%20Pharmacokinetics%20in%20Subjects%20with%20Mild-to-Moderate%20Alzhei

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each participant was to complete a 3-week placebo run-in period then receive a treatment sequence of either varenicline followed by placebo, or placebo followed by varenicline, separated by a 3-week placebo washout period. Of 92 participants screened, 66 participants were randomized to treatment.
Groups:
- Varenicline Then Placebo: Varenicline 0.5 mg once daily for 1 week followed by 0.5 mg twice daily (BID) for 1 week followed by 1 mg BID for 4 weeks; then placebo once daily for 1 week followed by placebo BID for 5 weeks.
- Placebo Then Varenicline: Placebo once daily for 1 week followed by placebo twice daily (BID) for 5 weeks; then varenicline 0.5 mg once daily for 1 week followed by 0.5 mg BID for 1 week followed by 1 mg BID for 4 weeks.
Period: Period 1
Arm/Group | Varenicline Then Placebo | Placebo Then Varenicline
Started | 32 | 34
Treated | 31 | 33
Completed | 26 | 29
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Other | 0 | 2
Not completed — Adverse Event | 4 | 0
Not completed — Randomized but not Treated | 1 | 1
Period: Placebo Washout
Arm/Group | Varenicline Then Placebo | Placebo Then Varenicline
Started | 26 | 29
Completed | 26 | 29
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Varenicline Then Placebo | Placebo Then Varenicline
Started | 26 | 29
Completed | 26 | 28
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Then Varenicline: Placebo twice a day (BID) initiated with a 2-week titration regimen (Week 1: once a day [QD]; Week 2: BID), followed by varenicline 1 mg BID initiated with a 2-week titration regimen (Week 1: 0.5 mg QD; Week 2: 0.5 mg BID).
- Total: Total of all reporting groups
Arm/Group | Varenicline Then Placebo | Placebo Then Varenicline | Total
Number analyzed (Participants) | 32 | 34 | 66
Age Continuous [Mean (Standard Deviation); unit: years] | 71.5 (8.7) | 73.9 (5.8) | 72.7 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Alzheimer's Disease Assessment Scale-Cognitive Subscale 75 (ADAS-Cog 75) at Week 6
Description: 12-item scale to assess severity of cognitive impairment in AD. Items include word recall, naming objects and fingers, following commands, constructional praxis, ideational praxis, orientation, word recognition, spoken language ability, comprehension of spoken language, word finding difficulty in spontaneous speech, remembering test instructions, and concentration/distractibility. Total score range from 0-75 with 75 indicating worse cognition.
Time Frame: Week 6
Population: Full analysis set (FAS): all participants who were randomized and took at least 1 dose of randomized study medication. N = number of participants with ADAS-Cog 75 results at Week 6.
Measure: Least Squares Mean (Standard Error); unit: units on scale
Groups:
- Varenicline: Varenicline 0.5 mg once daily for 1 week followed by 0.5 mg twice daily (BID) for 1 week followed by 1 mg BID for 4 weeks.
- Placebo: Placebo once daily for 1 week followed by placebo twice daily (BID) for 5 weeks.
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 53 | 55
units on scale | 18.07 (0.942) | 18.49 (0.939)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Difference from placebo. Analyzed using a mixed effects longitudinal linear model with subject (nested within sequence) as a random effect and fixed effects stratum, site, period, sequence, treatment, week, and treatment by week; Test type: Superiority or Other; p = 0.3873, ANCOVA — ANCOVA model using unstructured covariance structure; Type I error rate for primary hypothesis was 5%; no adjustments made for multiplicity; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.37 to 0.53]

2. Secondary Outcome: Alzheimer's Disease Assessment Scale-Cognitive Subscale 75 (ADAS-Cog 75) at Week 3
Description: as for outcome 1
Time Frame: Week 3
Population: FAS; N = number of participants with ADAS-Cog 75 results at Week 3.
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 58 | 54
units on scale | 19.87 (0.935) | 19.31 (0.941)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2465, ANCOVA — ANCOVA model using unstructured covariance structure; tested using a nominal 5% Type I error rate; no adjustments made for multiplicity; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [-0.39 to 1.49]

3. Secondary Outcome: Alzheimer's Disease Assessment Scale-Cognitive Subscale 70 (ADAS-Cog 70) at Week 3
Description: 11-item scale designed to assess the severity of cognitive impairments in AD subjects. Items include word recall, naming objects and fingers, following commands, constructional praxis, ideational praxis, orientation, word recognition, spoken language ability, comprehension of spoken language, word finding difficulty in spontaneous speech, and remembering test instructions. Total score range from 0-70 with 70 indicating worse cognition.
Time Frame: Week 3
Population: FAS. N = number of participants with ADAS-Cog 70 results at Week 3.
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 58 | 54
units on scale | 19.60 (0.880) | 19.01 (0.885)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Difference from placebo analyzed using a mixed effects longitudinal linear model with subject (nested within sequence) as a random effect and fixed effects stratum, site, period, sequence, treatment, week, and treatment by week; Test type: Superiority or Other; p = 0.2092, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [-0.33 to 1.50]

4. Secondary Outcome: Alzheimer's Disease Assessment Scale-Cognitive Subscale 70 (ADAS-Cog 70) at Week 6
Description: as for outcome 3
Time Frame: Week 6
Population: FAS. N = number of participants with ADAS-Cog 70 results at Week 6.
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 53 | 55
units on scale | 17.86 (0.886) | 18.23 (0.884)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.4339, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-1.30 to 0.56]

5. Secondary Outcome: Mean Clinical Global Impression - Improvement (CGI-I) Score at Week 6
Description: CGI-I: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected.
Time Frame: Week 6
Population: FAS; N = number of participants with a CGI-I score at Week 6.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 54 | 55
units on a scale | 3.71 (0.103) | 3.70 (0.102)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Difference from placebo analyzed using a mixed effects linear model with subject (nested within sequence) as a random effect, and stratum, site, period, sequence, and treatment as fixed effects; Test type: Superiority or Other; p = 0.9745, ANCOVA; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.26 to 0.27]

6. Secondary Outcome: Neuropsychiatric Inventory (NPI) Total Score at Week 3
Description: Caregiver interview-based rating scale assessing 12 behavioral disturbances occurring in dementia: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, appetite/eating, and sleep. Each symptom score derived by frequency of symptoms * severity of symptoms (range 0-12). Total score = sum of symptom scores; range: 0-144 with higher score indicating greater behavioral disturbances.
Time Frame: Week 3
Population: FAS. N = number of participants with a NPI total score at Week 3.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 59 | 54
scores on scale | 2.97 (0.845) | 2.29 (0.858)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2852, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.68, 95% CI 2-sided [-0.57 to 1.92]

7. Secondary Outcome: Neuropsychiatric Inventory (NPI) Total Score at Week 6
Description: as for outcome 6
Time Frame: Week 6
Population: FAS. N = number of participants with a NPI total score at Week 6.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 54 | 55
scores on scale | 3.82 (0.857) | 2.55 (0.855)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0468, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.28, 95% CI 2-sided [0.02 to 2.53]

8. Secondary Outcome: Computerized Test Battery for Cognition (CogState) Tasks: Detection at Week 1
Description: Assessment of the cognitive domain psychomotor function through yes or no responses within 5 minutes to 30 trials; score range: 0 to 3.69. Performance variable: speed of performance; average of the log10 t transformed reaction time for correct responses. Reaction times longer than 5 seconds (log10 [5000]) were excluded as reflecting responses that were abnormally slow.
Time Frame: Week 1
Population: FAS; N = number of participants with a CogState score for Detection at Week 1.
Measure: Least Squares Mean (Standard Error); unit: log10 millisecond
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 59 | 56
log10 millisecond | 2.65 (0.015) | 2.64 (0.015)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8811, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.02 to 0.03]

9. Secondary Outcome: Computerized Test Battery for Cognition (CogState) Tasks: Detection at Week 3
Description: as for outcome 8
Time Frame: Week 3
Population: FAS; N = number of participants with a CogState score for Detection at Week 3.
Measure: Least Squares Mean (Standard Error); unit: log10 millisecond
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 58 | 54
log10 millisecond | 2.65 (0.015) | 2.63 (0.015)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0830, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.00 to 0.05]

10. Secondary Outcome: Computerized Test Battery for Cognition (CogState) Tasks: Detection at Week 6
Description: as for outcome 8
Time Frame: Week 6
Population: FAS; N = number of participants with a CogState score for Detection at Week 6.
Measure: Least Squares Mean (Standard Error); unit: log10 millisecond
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 53 | 55
log10 millisecond | 2.64 (0.015) | 2.65 (0.015)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.7226, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.03 to 0.02]

11. Secondary Outcome: Computerized Test Battery for Cognition (CogState) Tasks: Continuous Paired Associate Learning (CPAL) at Week 1
Description: Assessment of the cognitive domain visual episodic memory (associate learning) through responses within 7 minutes to 4 targets x 4 rounds (mild AD) or 3 targets x 4 rounds (moderate AD); score range: 35 to 100. Performance variable: number of errors made in correctly placing each of the 4 patterns in their location four times.
Time Frame: Week 1
Population: FAS; N = number of participants with a CogState score for Continuous Paired Associate Learning at Week 1.
Measure: Least Squares Mean (Standard Error); unit: errors
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 59 | 56
errors | 38.52 (2.586) | 40.05 (2.626)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Week 1: difference from placebo. Analyzed using a mixed effects longitudinal linear model with subject (nested within sequence) as a random effect and fixed effects stratum, site, period, sequence, treatment, week, and treatment by week; Test type: Superiority or Other; p = 0.5588, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.53, 95% CI 2-sided [-6.68 to 3.62]

12. Secondary Outcome: Computerized Test Battery for Cognition (CogState) Tasks: Continuous Paired Associate Learning (CPAL) at Week 3
Description: as for outcome 11
Time Frame: Week 3
Population: FAS; N = number of participants with a CogState score for Continuous Paired Associate Learning at Week 3.
Measure: Least Squares Mean (Standard Error); unit: errors
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 58 | 54
errors | 39.43 (2.600) | 43.57 (2.656)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.1173, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -4.15, 95% CI 2-sided [-9.34 to 1.05]

13. Secondary Outcome: Computerized Test Battery for Cognition (CogState) Tasks: Continuous Paired Associate Learning (CPAL) at Week 6
Description: as for outcome 11
Time Frame: Week 6
Population: FAS; N = number of participants with a CogState score for Continuous Paired Associate Learning at Week 6.
Measure: Least Squares Mean (Standard Error); unit: errors
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 53 | 55
errors | 41.67 (2.668) | 42.98 (2.641)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.6251, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.31, 95% CI 2-sided [-6.58 to 3.96]

14. Secondary Outcome: Computerized Test Battery for Cognition (CogState) Tasks: One Back Working Memory at Week 1
Description: Assessment of the cognitive domain working memory through yes or no responses to 30 trials within 5 minutes; score range: 0 to 1.57. Performance variable: accuracy of performance; arcsine transformation of proportion correct responses.
Time Frame: Week 1
Population: FAS; N = number of participants with a CogState score for One Back Working Memory at Week 1.
Measure: Least Squares Mean (Standard Error); unit: arcsine proportion correct
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 59 | 56
arcsine proportion correct | 0.94 (0.031) | 0.94 (0.031)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.9109, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.05 to 0.05]

15. Secondary Outcome: Computerized Test Battery for Cognition (CogState) Tasks: One Back Working Memory at Week 3
Description: as for outcome 14
Time Frame: Week 3
Population: FAS; N = number of participants with a CogState score for One Back Working Memory at Week 3.
Measure: Least Squares Mean (Standard Error); unit: arcsine proportion correct
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 58 | 54
arcsine proportion correct | 0.96 (0.031) | 0.97 (0.032)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.6632, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.06 to 0.04]

16. Secondary Outcome: Computerized Test Battery for Cognition (CogState) Tasks: One Back Working Memory at Week 6
Description: as for outcome 14
Time Frame: Week 6
Population: FAS; N = number of participants with a CogState score for One Back Working Memory at Week 6.
Measure: Least Squares Mean (Standard Error); unit: arcsine proportion correct
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 53 | 55
arcsine proportion correct | 0.95 (0.032) | 0.96 (0.031)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.5450, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.07 to 0.04]

17. Secondary Outcome: Computerized Test Battery for Cognition (CogState) Tasks: Visual Learning at Week 1
Description: Assessment of the cognitive domain episodic memory through yes or no responses within 5 minutes to 4 targets repeated among 6 distractors on 4 rounds (mild Alzheimer's disease [AD], or 3 targets repeated among 4 distractors on 4 rounds (moderate AD) ; score range: 0 to 1.57. Performance variable: accuracy of performance; arcsine transformation of proportion correct responses.
Time Frame: Week 1
Population: FAS; N = number of participants with a CogState score for Visual Learning at Week 1.
Measure: Least Squares Mean (Standard Error); unit: arcsine proportion correct
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 59 | 56
arcsine proportion correct | 0.83 (0.015) | 0.81 (0.016)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2799, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.02 to 0.05]

18. Secondary Outcome: Computerized Test Battery for Cognition (CogState) Tasks: Visual Learning at Week 3
Description: as for outcome 17
Time Frame: Week 3
Population: FAS; N = number of participants with a CogState score for Visual Learning at Week 3.
Measure: Least Squares Mean (Standard Error); unit: arcsine proportion correct
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 58 | 54
arcsine proportion correct | 0.82 (0.016) | 0.82 (0.016)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Difference from placebo aAnalyzed using a mixed effects longitudinal linear model with subject (nested within sequence) as a random effect and fixed effects stratum, site, period, sequence, treatment, week, and treatment by week; Test type: Superiority or Other; p = 0.9675, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.03 to 0.04]

19. Secondary Outcome: Computerized Test Battery for Cognition (CogState) Tasks: Visual Learning at Week 6
Description: as for outcome 17
Time Frame: Week 6
Population: FAS; N = number of participants with a CogState score for Visual Learning at Week 6.
Measure: Least Squares Mean (Standard Error); unit: arcsine proportion correct
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 53 | 55
arcsine proportion correct | 0.83 (0.016) | 0.84 (0.016)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.5008, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.05 to 0.02]

20. Secondary Outcome: Computerized Test Battery for Cognition (CogState) Tasks: Identification at Week 1
Description: Assessment of the cognitive domain visual attention through a yes or no response to 30 trials within 5 minutes; score range: 0 to 3.69. Performance variable: speed of performance; average log10 transformed reaction time for correct responses. Reaction times longer than 5 seconds ( log10 [5000]) were excluded as reflecting responses that were abnormally slow.
Time Frame: Week 1
Population: FAS; N = number of participants with a CogState score for Identification at Week 1.
Measure: Least Squares Mean (Standard Error); unit: log10 millisecond
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 59 | 56
log10 millisecond | 2.79 (0.011) | 2.80 (0.011)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2245, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.03 to 0.01]

21. Secondary Outcome: Computerized Test Battery for Cognition (CogState) Tasks: Identification at Week 3
Description: as for outcome 20
Time Frame: Week 3
Population: FAS; N = number of participants with a CogState score for Identification at Week 3.
Measure: Least Squares Mean (Standard Error); unit: log10 millisecond
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 58 | 54
log10 millisecond | 2.79 (0.011) | 2.80 (0.011)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.4974, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.03 to 0.01]

22. Secondary Outcome: Computerized Test Battery for Cognition (CogState) Tasks: Identification at Week 6
Description: as for outcome 20
Time Frame: Week 6
Population: FAS; N = number of participants with a CogState score for Identification at Week 6.
Measure: Least Squares Mean (Standard Error); unit: log10 millisecond
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 52 | 55
log10 millisecond | 2.79 (0.012) | 2.79 (0.011)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8525, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.02 to 0.02]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 2/60 | 0/59
Other Adverse Events (participants affected / at risk) | 56/60 | 37/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=60) | Placebo (N=59)
Asthenia (General disorders) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=60) | Placebo (N=59)
External ear inflammation (Ear and labyrinth disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Cataract (Eye disorders) | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Eye disorder (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 1
Gastric disorder (Gastrointestinal disorders) | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 17 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 12 | 0
Asthenia (General disorders) | 2 | 1
Fatigue (General disorders) | 2 | 1
Feeling abnormal (General disorders) | 1 | 1
Hunger (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Urine analysis abnormal (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 1
White blood cells urine positive (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 13 | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 8 | 0
Headache (Nervous system disorders) | 7 | 4
Intention tremor (Nervous system disorders) | 1 | 1
Lethargy (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Depressed mood (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Sleep disorder (Psychiatric disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 2 | 0
Intermittent claudication (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.